CLINICAL TRIAL: NCT04673929
Title: Transoral Robotic Surgery for rECurrent Tumours of the Upper Aerodigestive Tract
Acronym: RECUT
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5156
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Recurrent Head and Neck Cancer
Keywords: Recurrent head and neck cancer; transoral robotic surgery; TORS; HNC recurrence
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with Head & Neck Cancer recurrence treated with Transoral Robotic Surgery: Report of disease-free survival at 2 years for patients with Head & Neck Cancer recurrence treated with Transoral Robotic Surgery

SUMMARY:
transoral Robotic surgery for rECurrent tumours of the Upper aerodigestive Tract

DETAILED DESCRIPTION:
Head and neck cancer (HNC) is the 6th most common type of cancer in the world and is increasing in incidence. Squamous cell carcinomas (SCC) account for the majority of these HNCs. An increasing number of these SCCs are being found to be associated with the Human Papilloma Virus (HPV) which has also been shown to be associated with a more favourable outcome. These HPV related cancers tend to affect younger patients with fewer comorbidities. As such, we are finding a larger cohort of patients are surviving for longer after treatment for their primary cancers.

HNC patients are over 11 times more likely to experience a second head and neck primary cancer than the general population over 20 years of follow up (SIR 11.2, 95% CI [10.6-11.8]). In addition to second primaries, patients may suffer from residual disease after treatment for their initial primary, identified within a 12 month period, or recurrent disease, cancer at the same site identified within 5 years. Treatment for all of these cancers, which we will broadly term 'recurrent' cancers for the purposes of this study, can be complex. Commonly, radiotherapy will have formed part of the treatment regime at either the primary site or to the neck for these patients. Radiotherapy causes fibrosis in the irradiated tissues, reducing tissue pliability, contributing to trismus and reducing healing potential at the effected sites. This can pose significant challenges to any further surgical intervention, which may form the mainstay of any subsequent management if re-irradiation is not an option or not indicated. Surgery must then look to be as minimally invasive as possible in order to maximise functional outcomes and reduce disruption of affected tissues.

Options for surgery have traditionally involved transmandibular and transcervical routes. More recently transoral routes have been adopted as endoscopic instruments become more widely available and adopted. Transoral Robotic Surgery (TORS) is the latest development in the field which confers some significant advantages to the surgeon and to the patient. For the surgeon, the endoscopic view is binocular, giving a close objective lens and excellent depth perception. Further, the instruments have wrists which sit within the body cavity, allowing manipulation of the tissues beyond the direct line of sight through the oral stoma. For the patient, there is less disrupted tissue if access incisions are avoided, reducing the volume of tissue that would be susceptible to scarring which can affect swallowing function or lead to fistula formation.

However, there are little data to show oncological and functional outcomes are acceptable following TORS surgery for recurrent cancers. This is in part as it is a relatively new technology and in part because whilst increasingly common, the absolute number of surgeries performed remains relatively low at individual centres. Published outcomes have shown 2 year disease-free survival rates around 75%. The RECUT study aims to use a collaborative methodology to document the outcomes from TORS for recurrent HNC being performed at a number of high volume centres across the globe.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18
* Previous Head & Neck Cancer treated with radiotherapy
* Undergoing Transoral Robotic Surgery as part of their management for recurrent disease
* Surgery performed on or before July 31st 2018.

Exclusion Criteria:

* Transoral Robotic Surgery used in a diagnostic setting only
* Nasopharyngeal and thyroid cancers

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals aged over 18 with previous Head and Neck Cancer treated with radiotherapy and undergoing Transoral Robotic Surgery as part of their management for recurrent disease. Surgery performed on or before July 31st 2018.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Head and Neck Unit, Royal Marsden Hospital, London, Greater London
  - Royal Marsden Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Shield KD, Ferlay J, Jemal A, Sankaranarayanan R, Chaturvedi AK, Bray F, Soerjomataram I. The global incidence of lip, oral cavity, and pharyngeal cancers by subsite in 2012. CA Cancer J Clin. 2017 Jan;67(1):51-64. doi: 10.3322/caac.21384. Epub 2016 Oct 19. PMID 28076666
- [Background] INTEGRATE (The National ENT Trainee Research Network). British Association of Head and Neck Oncologists Surveillance audit 2018. Unpublished
- [Background] Chuang SC, Scelo G, Tonita JM, Tamaro S, Jonasson JG, Kliewer EV, Hemminki K, Weiderpass E, Pukkala E, Tracey E, Friis S, Pompe-Kirn V, Brewster DH, Martos C, Chia KS, Boffetta P, Brennan P, Hashibe M. Risk of second primary cancer among patients with head and neck cancers: A pooled analysis of 13 cancer registries. Int J Cancer. 2008 Nov 15;123(10):2390-6. doi: 10.1002/ijc.23798. PMID 18729183
- [Background] Gross ND, Hanna EY. The Role of Surgery in the Management of Recurrent Oropharyngeal Cancer. Recent Results Cancer Res. 2017;206:197-205. doi: 10.1007/978-3-319-43580-0_15. PMID 27699540
- [Background] Paleri V, Fox H, Coward S, Ragbir M, McQueen A, Ahmed O, Meikle D, Saleh D, O'Hara J, Robinson M. Transoral robotic surgery for residual and recurrent oropharyngeal cancers: Exploratory study of surgical innovation using the IDEAL framework for early-phase surgical studies. Head Neck. 2018 Mar;40(3):512-525. doi: 10.1002/hed.25032. Epub 2017 Dec 15. PMID 29244229
- [Background] Hamilton D, Paleri V. Role of transoral robotic surgery in current head & neck practice. Surgeon. 2017 Jun;15(3):147-154. doi: 10.1016/j.surge.2016.09.004. Epub 2016 Oct 11. PMID 27742406
- [Background] Weinstein GS, O'Malley BW Jr, Cohen MA, Quon H. Transoral robotic surgery for advanced oropharyngeal carcinoma. Arch Otolaryngol Head Neck Surg. 2010 Nov;136(11):1079-85. doi: 10.1001/archoto.2010.191. PMID 21079160
- [Background] White H, Ford S, Bush B, Holsinger FC, Moore E, Ghanem T, Carroll W, Rosenthal E, Sweeny L, Magnuson JS. Salvage surgery for recurrent cancers of the oropharynx: comparing TORS with standard open surgical approaches. JAMA Otolaryngol Head Neck Surg. 2013 Aug 1;139(8):773-8. doi: 10.1001/jamaoto.2013.3866. PMID 23949352
- [Background] Dabas S, Dewan A, Ranjan R, Dewan AK, Shukla H, Sinha R. Salvage Transoral Robotic Surgery for Recurrent or Residual Head and Neck Squamous Cell Carcinoma: A Single Institution Experience. Asian Pac J Cancer Prev. 2015;16(17):7627-32. doi: 10.7314/apjcp.2015.16.17.7627. PMID 26625773
- [Background] Piccirillo JF. Importance of comorbidity in head and neck cancer. Laryngoscope. 2000 Apr;110(4):593-602. doi: 10.1097/00005537-200004000-00011. PMID 10764003
- [Background] Paleri V, Wight RG. Applicability of the adult comorbidity evaluation - 27 and the Charlson indexes to assess comorbidity by notes extraction in a cohort of United Kingdom patients with head and neck cancer: a retrospective study. J Laryngol Otol. 2002 Mar;116(3):200-5. doi: 10.1258/0022215021910528. PMID 11893262
- [Background] Microsoft. Excel for Mac [Internet]. Redmond, Washington, USA: Microsoft Corporation; 2018. Available from: https://products.office.com/
- [Background] R Core Team. R: A language and environment for statistical computing [Internet]. Vienna, Austria: R Foundation for Statistical Computing; 2013. Available from: http://www.R-project.org/
- [Background] RStudio Team. RStudio: Integrated Development Environment for R [Internet]. Boston, MA: RStudio, Inc.; 2015. Available from: http://www.rstudio.com/
- [Background] ICMJE | Recommendations | Defining the Role of Authors and Contributors [Internet]. [cited 2019 Jan 23];Available from: http://www.icmje.org/recommendations/browse/roles-and-responsibilities/defining-the-role-of-authors-and-contributors.html
- [Derived] Hardman JC, Holsinger FC, Brady GC, Beharry A, Bonifer AT, D'Andrea G, Dabas SK, de Almeida JR, Duvvuri U, Floros P, Ghanem TA, Gorphe P, Gross ND, Hamilton D, Kurukulasuriya C, Larsen MHH, Lin DJ, Magnuson JS, Meulemans J, Miles BA, Moore EJ, Pantvaidya G, Roof S, Rubek N, Simon C, Subash A, Topf MC, Van Abel KM, Vander Poorten V, Walgama ES, Greenlay E, Potts L, Balaji A, Starmer HM, Stephen S, Roe J, Harrington K, Paleri V. Transoral Robotic Surgery for Recurrent Tumors of the Upper Aerodigestive Tract (RECUT): An International Cohort Study. J Natl Cancer Inst. 2022 Oct 6;114(10):1400-1409. doi: 10.1093/jnci/djac130. PMID 35944904

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Head & Neck Cancer (HNC) Recurrence Treated With Transoral Robotic Surgery (TORS): Report of disease-free survival at 2 years for patients with HNC recurrence treated with TORS
Period: Overall Study
Arm/Group | Patients With Head & Neck Cancer (HNC) Recurrence Treated With Transoral Robotic Surgery (TORS)
Started | 278
Completed | 162
Not Completed | 116
Not completed — Death | 73
Not completed — Did not reach the 2 year follow up point (observational study) | 43

BASELINE CHARACTERISTICS:
Groups:
- Patients With HNC Recurrence Treated With TORS: Report of disease-free survival at 2 years for patients with HNC recurrence treated with TORS
Arm/Group | Patients With HNC Recurrence Treated With TORS
Number analyzed (Participants) | 278
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 166
  >=65 years | 112
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [56 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 222
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 278
Performance Status Scale - Head and Neck Normalcy of diet [Mean (Full Range); unit: units on a scale] — Normalcy of diet, public eating and understandability of speech assessed through interview, each scoring between 0 and 100.
  0 = Never understandable / Always eats alone/ Non-oral feeding 100 = No restrictions / always understandable
  units on a scale | 77.1 [0 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival at 2 Years
Description: Disease-free survival measured at 2 years for all recruited participants - data retrieved from medical records retrospectively
  Measured as 2 years post TORS procedure
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With HNC Recurrence Treated With TORS
Number analyzed (Participants) | 235
Participants | 111

2. Secondary Outcome: Overall Survival at 2 Years
Description: Overall survival at 2 years - number of living participants at end of 2 year follow up - data retrieved from medical records retrospectively
  Measured as 2 years post TORS procedure
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Head & Neck Cancer Recurrence Treated With Transoral Robotic Surgery: Report of survival at 2 years for patients with Head & Neck Cancer recurrence treated with Transoral Robotic Surgery
Arm/Group | Patients With Head & Neck Cancer Recurrence Treated With Transoral Robotic Surgery
Number analyzed (Participants) | 278
Participants | 192

3. Secondary Outcome: Rate of Gastrostomy Use at 1 Year
Description: Rate of gastrostomy use at 1 year - number of participants having a gastrostomy post surgery
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Head & Neck Cancer Recurrence Treated With Transoral Robotic Surgery: Report of gastrostomy use for patients with Head & Neck Cancer recurrence treated with Transoral Robotic Surgery
Arm/Group | Patients With Head & Neck Cancer Recurrence Treated With Transoral Robotic Surgery
Number analyzed (Participants) | 278
Participants | 109

4. Secondary Outcome: Rate of Tracheostomy Use at 1 Year
Description: Rate of tracheostomy use at 1 year
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Patients With Head & Neck Cancer Recurrence Treated With Transoral Robotic Surgery: Report of tracheostomy use for patients with Head & Neck Cancer recurrence treated with Transoral Robotic Surgery
Arm/Group | Patients With Head & Neck Cancer Recurrence Treated With Transoral Robotic Surgery
Number analyzed (Participants) | 277
Participants | 105

5. Primary Outcome: Disease-specific Survival at 2 Years
Description: Disease-specific survival measured at 2 years for all recruited participants - data retrieved from medical records retrospectively
  Measured as 2 years post TORS procedure
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With HNC Recurrence Treated With TORS
Number analyzed (Participants) | 278
Participants | 219

ADVERSE EVENTS:
Time Frame: Deaths recorded up to 5 years post TORS procedure - data collected retrospectively from medical records
Description: Deaths reported as adverse events, no other adverse event data collected
Arm/Group | Patients With HNC Recurrence Treated With TORS
All-Cause Mortality (participants affected / at risk) | 115/278
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT04673929/Prot_SAP_001.pdf